CLINICAL TRIAL: NCT01775332
Title: Interdisciplinary Pituitary Disorders Centre of Excellence: Assessment of Patient Education Tools
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMHAIF - 058
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Pituitary Neoplasms; Prolactinoma; ACTH-Secreting Pituitary Adenoma; Gigantism; Growth Hormone-Secreting Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms; Prolactinoma; ACTH-Secreting Pituitary Adenoma; Gigantism; Growth Hormone-Secreting Pituitary Adenoma | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention (Experimental): Educational Intervention - Access to educational materials provided (i.e. website, videos, brochure)
  Interventions: Other: Educational Intervention
- No Intervention/Use of Own Resources (No Intervention): No educational materials are provided to participants, but they can use their own resources

INTERVENTIONS:
Other: Educational Intervention — A brochure and access to a website including videos that contain detailed information about pituitary disorders will serve as the educational intervention.
  Arms: Educational Intervention

SUMMARY:
The purpose of this research study is to determine the utility of educational materials designed to inform patients of their pituitary condition, in an effort to assist the patients, families, and staff deal with pituitary tumours and related conditions in the best way possible. We have developed a website, informational videos, and a brochure for pituitary tumour patients and their families. The primary outcome measures will be 1) the level of knowledge that patients have of their condition before and after reviewing the materials provided; and 2) ease of use and user satisfaction of the materials. We hypothesize that our informative multimedia educational package will not only improve the health literacy and self-efficacy of patients and their families, but will also improve quality of care.

DETAILED DESCRIPTION:
This study involves a formative evaluation of the health literacy resources that we have already developed. We see approximately 60 new patients a year with pituitary disorders, plus the follow-up patients: all of these patients will be offered the opportunity to participate in the study. These materials include a website (containing videos, illustrations and written materials) and plain language educational brochures. The educational materials include information that patients will need throughout their experience with a pituitary tumour, ranging from the signs and symptoms of tumours, to long-term post-operative lifestyle changes. This evaluation will be a mixed-methods evaluation.

Part A (Think aloud) will use "think-aloud" processes to evaluate the usefulness and ease of use of a website that we have developed with patients and their families.

Part B (Resource assessment) will involve the use of questionnaires followed by semi-structured interviews with patients and families before and after using the resources.

ELIGIBILITY:
Inclusion Criteria:

* age equal to or greater than 18 years;
* capable of providing consent to participate on their own behalf;
* diagnosed with a pituitary disorder OR have a history of pituitary disorder AND a current/former patient at St. Michael's Hospital, OR be a caretaker of someone with a pituitary disorder;
* adequate written/verbal English skills.

Exclusion Criteria:

* Younger than 18 years;
* Unable to provide consent;
* Unable to communicate in written/verbal English, as all of the surveys and interviews are administered in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The level of knowledge that patients have of their condition before and after reviewing the materials provided, and ease of use of educational materials and user satisfaction | 1-2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cusimano, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Andrulis DP, Brach C. Integrating literacy, culture, and language to improve health care quality for diverse populations. Am J Health Behav. 2007 Sep-Oct;31 Suppl 1(Suppl 1):S122-33. doi: 10.5555/ajhb.2007.31.supp.S122. PMID 17931131
- [Background] Kan P, Cusimano M. Validation of a quality-of-life questionnaire for patients with pituitary adenoma. Can J Neurol Sci. 2006 Feb;33(1):80-5. doi: 10.1017/s0317167100004741. PMID 16583727
- [Background] Goguen, J. (2007). Perioperative management of the pituitary patients. Endocrinology Rounds, 7(9): 1-6. Retrieved February 2, 2011 from http://www.endocrinologyrounds.ca